CLINICAL TRIAL: NCT05071079
Title: A Clinical Study to Assess the Safety and Feasibility of Controlled Blood-stage Plasmodium Vivax Human Malaria Infection Through Experimental Inoculation of Cryopreserved Infected Erythrocytes in Healthy Thai Adults
Brief Title: A Controlled Human Vivax Malaria Infection Study Through Inoculation of Infected Erythrocytes
Acronym: MIST2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MAL21001
Record Dates: First submitted 2021-07-28; First posted 2021-10-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Plasmodium Vivax Infection
Keywords: controlled human malaria infection; Plasmodium Vivax Infection

STUDY DESIGN:
Intervention Model Description: Controlled Plasmodium vivax human malaria infection through experimental inoculation of cryopreserved infected erythrocytes in healthy Thai adults, with a randomized double blind design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded study; volunteers, clinical investigators, and study staff who perform laboratory study endpoint will be blinded to inoculation arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Challenge with whole dose blood-stage inoculum (neat) (Experimental): Whole dose: one whole vial, containing approximately 0.5 mL of red blood cells, will be reconstituted in 0.9% saline, to a total volume of 5 mL
  Interventions: Biological: An inoculum of malaria parasitised red blood cells with whole dose blood-stage inoculum
- Challenge with 1:5 dilution blood-stage inoculum (Experimental): 1:5 dilution: one fifth of a vial (containing approximately 0.1 mL of red blood cells) will be reconstituted in 0.9% saline, to a total volume of 5 mL.
  Interventions: Biological: An inoculum of malaria parasitised red blood cells with 1:5 dilution blood-stage inoculum
- Challenge with 1:10 dilution blood-stage inoculum (Experimental): 1:10 dilution: one tenth of a vial (containing approximately 0.05 mL of red blood cells) will be reconstituted in 0.9% saline, to a total volume of 5 mL.
  Interventions: Biological: An inoculum of malaria parasitised red blood cells with 1:10 dilution blood-stage inoculum
- Challenge with 1:20 dilution blood-stage inoculum (Experimental): 1:20 dilution: one twenties of a vial (containing approximately 0.025 mL of red blood cells) will be reconstituted in 0.9% saline, to a total volume of 5 mL.
  Interventions: Biological: An inoculum of malaria parasitised red blood cells with 1:20 dilution blood-stage inoculum

INTERVENTIONS:
Biological: An inoculum of malaria parasitised red blood cells with whole dose blood-stage inoculum — An inoculum of malaria parasitised red blood cells reconstituted in 0.9% normal saline, to a total volume of 5 mL; challenge with whole dose blood-stage inoculum (neat)
  Arms: Challenge with whole dose blood-stage inoculum (neat)
Biological: An inoculum of malaria parasitised red blood cells with 1:5 dilution blood-stage inoculum — An inoculum of malaria parasitised red blood cells reconstituted in 0.9% normal saline, to a total volume of 5 mL; challenge with 1:5 dilution blood-stage inoculum
  Arms: Challenge with 1:5 dilution blood-stage inoculum
Biological: An inoculum of malaria parasitised red blood cells with 1:10 dilution blood-stage inoculum — An inoculum of malaria parasitised red blood cells reconstituted in 0.9% normal saline, to a total volume of 5 mL; challenge with 1:10 dilution blood-stage inoculum
  Arms: Challenge with 1:10 dilution blood-stage inoculum
Biological: An inoculum of malaria parasitised red blood cells with 1:20 dilution blood-stage inoculum — An inoculum of malaria parasitised red blood cells reconstituted in 0.9% normal saline, to a total volume of 5 mL; challenge with 1:20 dilution blood-stage inoculum
  Arms: Challenge with 1:20 dilution blood-stage inoculum

SUMMARY:
The primary objectives of this study are to assess the safety and feasibility of blood-stage controlled human P. vivax malaria infection (CHMI) in healthy adult Thai volunteers through experimental injection of cryopreserved P. vivax infected erythrocytes, and to choose the optimal inoculation dose for future P. vivax CHMI studies. In this study, blood-stage CHMI will be conducted in 8 volunteers per inoculum stock who will each be infected with P. vivax by experimental injection with cryopreserved P. vivax infected erythrocytes, which were collected from the controlled human Plasmodium vivax malaria infection model through experimental sporozoite infection in Thai adults (NCT04083508) . There are currently 4 stocks of inocula from 6 volunteers in the NCT04083508 study, which have differing quantities and stages of parasites.

The total number of volunteers of this study will be up to 48 (8 volunteers per inocula stock). The volunteers will be monitored closely as in-patients in the Hospital for Tropical Diseases, and will be treated according to the Research Proposal.

This study is funded by the UK Wellcome Trust. The grant reference number are Oxford/MORU: 212336/Z/18/Z and 212336/Z/18/A, and Mahidol University: 212336/A/18/Z and 212336/A/18/A.

DETAILED DESCRIPTION:
This study is a blood-stage P. vivax human challenge study with the primary aim of assessing the safety and feasibility of a challenge model using banks of cryopreserved P. vivax infected erythrocytes produced from NCT04083508 study to identify the dose of the inocula to be used in the future CHMI studies.

Forty-eight healthy Thai adults, aged between 20 and 55 years will be recruited at the Clinical Therapeutics Unit (CTU) in the Hospital for Tropical Diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok. The overall period of each volunteer's participation will be 13 months: 2-week screening process prior to the Day 0 challenge, about 2-week inoculum process until reaching malarial treatment criteria, and follow-up period for 1 year after malarial treatment. All inclusion and exclusion criteria will be checked to ensure eligibility criteria have been met prior to Day 0.

Volunteers will be admitted to the hospital one day prior to challenged day. All eligible volunteers will have physical examinations. Serum pregnancy test (women only), malaria diagnosis, complete blood count (CBC), and biochemistry will be tested. Glucose -6-phospate dehydrogenase (G6PD) test and malaria immunological profiles will be tested for baseline information.

On the challenged day (Day 0), four different doses of inoculum (one whole vial,1:5 dilution, 1:10 dilution, and 1:20 dilution) will be assessed. Each dose of inoculum will be tested in 2 volunteers to identify the lowest concentration producing a reliable infection within a practicable timeframe. Therefore, there will be 8 volunteers enrolled per inoculum bank.

The assessment will be repeated in each inoculum bank. There are currently 4 inoculum banks and 20 volunteers have been enrolled to date so 28 volunteers will be enrolled into this study.

From Day 1 after challenge, the volunteers will be assessed once daily until malaria qPCR becomes positive. The assessment includes a clinical well-being check, physical examination, vital signs, and blood drawn for parasitaemia (malaria blood film, qPCR, and gametocyte qPCR) and membrane feeding to assess the transmissibility of gametocyte. Malaria immunology and CBC will be performed on day 4 and the day that qPCR become positive.

After qPCR becomes positive the monitoring of clinical well-being will continue. Blood will be drawn twice daily to monitor blood parasitaemia and allow membrane feeding to assess the transmissibility of gametocyte. Malaria immunology, CBC, and blood biochemistry will be performed on day that volunteer reach malaria treatment criteria.

When the malaria slide positivity and/or symptoms thresholds have been reached study physician will immediately prescribe antimalarial treatment with chloroquine according to local standard guidelines. Blood will be collected to test for malaria (blood films and qPCR) once daily until clinically recovered and two consecutive malaria blood films are negative (completing of the chloroquine treatment course) and volunteers will be discharged from the hospital. Before discharge from the hospital, HIV-I and HIV-II antigen, HBV and HCV serology, COVID-19 testing (RT-PCR) and COVID-19 serology test will be carried out to confirm that volunteers did not acquire COVID-19 during their inpatient stay.

If any volunteer reaches day 21 post-challenge without a positive malaria blood film, they shall be started on 3-day course of antimalarial treatment (chloroquine).

If a volunteer withdraws/is withdrawn from the study after challenge but before reaching the criteria for malaria treatment, then a complete, appropriate, curative course of antimalarial therapy must be completed

After discharge from the hospital, there will be out-patient visits on day 7, 28, 60, 90, 180, and 1 year post antimalarial treatment initiation. Blood will be collected to detect malaria parasites by blood film and qPCR, and for malaria gametocyte qPCR, membrane feeding assays (MFA), HIV-I and HIV-II antigen, HBV, HCV, CMV, and EBV, malaria immune response, CBC, and biochemistry according to the study protocol.

Data analysis

The safety of the CHMI will be assessed by descriptive analysis of the frequency, incidence and nature of adverse events and serious adverse events arising during the study. Since this is a feasibility study conducted in 2 volunteers per dosing group, formal statistical hypothesis testing will not be used for most analyses due to the limited sample size, and only a brief Statistical Analysis Plan (SAP) will be developed and finalized prior to database lock.

The study will be conducted in accordance with the current approved protocol, the International Conference on Harmonisation-Good Clinical Practice (ICH GCP), relevant regulations, and standard operating procedures. Data will be evaluated for compliance with the protocol and accuracy in relation to source documents. Following written standard operating procedures, the monitors will verify that the clinical study is conducted and data are generated, documented and reported in compliance with the protocol.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must meet all of the following criteria to be eligible for the study:

1. Healthy Thai adult aged 20 to 55 years with weight at least 50 kg.
2. Red blood cells positive for the Duffy antigen/chemokine receptor (DARC)
3. Women only: Must practice continuous effective contraception for the duration of study period until 3 months post-challenge.
4. COVID-19 vaccination at least two doses of COVID-19 vaccines approved by WHO.
5. Agreement to refrain from blood donation during the course of the study and for 1 year after the initiation of antimalarial treatment.
6. Willing to be admitted in the Hospital for Tropical Diseases for clinical monitoring, until antimalarial treatment is completed and their symptoms are settling.
7. Willing to take a curative antimalarial treatment following CHMI.
8. Willing to reside in Bangkok and its vicinity for 2 months after malarial treatment initiation.
9. Able to read and write in Thai.
10. Provide written informed consent to participate in the trial
11. Answer all questions on the informed consent quiz correctly
12. Educational level: has at least an undergraduate degree

Exclusion Criteria:

The volunteer must NOT enter the study if any of the following apply:

1. Positive malaria qPCR OR malaria film
2. Presence of any medical condition (either physical or psychological) which in the judgment of the investigator would place the participant at undue risk or interfere with the results of the study (e.g. serious underlying cardiac, renal, hepatic or neurological disease; severe malnutrition; congenital defects or febrile condition)
3. Presence of chronic disease or chronically use of medication
4. Use of systemic antibiotics with known antimalarial activity in the 30 days before challenge (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)
5. Use of immunoglobulins or blood products (e.g. blood transfusion) at any time in the 1 year preceding enrolment
6. Receipt of an investigational product, any vaccine in the 30 days preceding enrolment (D0), or planned receipt during the study period
7. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data or the P. vivax parasite as assessed by the Investigator.
8. Any confirmed, or suspected immunosuppressive, or immunodeficient state, including HIV infection, asplenia, history of splenectomy, recurrent, severe infections, and chronic infection
9. Immunosuppressant medication within the past 6 months preceding enrolment (D0) (inhaled and topical steroids are allowed)
10. History of allergic disease or reactions likely to be exacerbated by malaria infection
11. Female participant who is pregnant as evidenced by positive beta-human chorionic gonadotropin (β-HCG) test, lactating, or planning pregnancy during the course of the study
12. Contraindications to the use of antimalarial treatment (e.g. chloroquine, atovaquone / proguanil or dihydroartemisinin/piperaquine)
13. Use of medications known to have a potentially clinically significant interaction with the antimalarial drug that will be used in this study (chloroquine, atovaquone / proguanil or dihydroartemisinin/piperaquine)
14. Known existing positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease
15. History of cardiac arrhythmia, including clinically relevant bradycardia
16. Family history of congenital QT prolongation or sudden death
17. Any clinical condition, including using medications, known to prolong the QT interval.
18. Screening electrocardiogram (ECG) demonstrates a QTc interval ≥ 450 ms.
19. Suspected or known or history of alcohol abuse
20. Suspected or known or history of drug abuse.
21. Concurrently participating in another clinical study, at any time during the study period
22. Haemoglobin < 11 g/dL
23. Positive hepatitis B surface antigen or seropositive for hepatitis C virus
24. Finding on safety laboratory values as defined below:

    * Abnormal AST (AST > 40 U/L for male, and > 32 U/L for female [upper normal range])
    * Abnormal ALT (ALT > 41 U/L for male, and > 33 U/L for female [upper normal range])
    * Abnormal serum creatinine (Scr) (Creatinine [Cr] > 1.17 mg/dL for male, and > 0.95 mg/dL for female [upper normal range])
    * Abnormalities corrected calcium and magnesium blood levels
25. Blood group Rhesus negative
26. Blood incompatibility to the inoculum
27. Positive for COVID-19 diagnosed by RT-PCR

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incident of treatment-emergent adverse events of blood-stage controlled human P. vivax malaria infection | Through study completion, over one year
  Measured by (serious) adverse event (AE) occurrences
Choosing the optimal inoculation dose for future P. vivax CHMI studies, which will be the lowest concentration that produces a reliable infection within a comparable timeframe as compare to the highest concentration. | Through study completion, over one year
  The optimal inoculation dose for future P. vivax CHMI studies, which will be the lowest concentration that produces a reliable infection within a comparable timeframe as compare to the highest concentration
Feasibility of primary P. vivax blood-stage CHMI, as measured by successful infection (development of detectable persistent parasitaemia by thick blood film +/- clinical symptoms) | Through study completion, over one year

SECONDARY OUTCOMES:
Geometric mean and standard deviation/error of Pvs25 gene transcript copy number/microL at each time point | Challenge day; day 1 to 5 or up to day of treatment and during subsequent days of follow-up through study completion, over one year
  Measured by qPCR in experimental P. vivax infection through blood-stage challenge
Transmissibility of gametocytes from the infected volunteer to Anopheles mosquito vector | Through study completion, over one year
  Measured by gametocytes from the infected volunteer to Anopheles mosquito vector using Membrane feeding assay
Cellular Immune response to primary P. vivax infection (frequencies, percentages (%), and expression level of mononuclear cells) | Day-1, Day 2, Day 5, Day of blood donation, DayRx7, DayRx28, DayRx90, DayRx1 year
  Immune cells including Innate and adaptive immune cells react and express during the PV infection (profile and frequency)
Level of antibodies and cytokines responses to primary P. vivax infection during different phase of infection | Day-1, Day 2, Day 5, Day of blood donation, DayRx7, DayRx28, DayRx90, DayRx1 year
  Immune cells defense PV antigen by determining the level of antibody response and inflammatory cytokine

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Day, MD, Principal Investigator — University of Oxford
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Volunteer's data and results from blood analyses stored in our database may be shared with other researchers to use in the future. However, the other researchers will not be given any information that could identify the subject.

REFERENCES:
- [Background] Baird JK. Evidence and implications of mortality associated with acute Plasmodium vivax malaria. Clin Microbiol Rev. 2013 Jan;26(1):36-57. doi: 10.1128/CMR.00074-12. PMID 23297258
- [Background] Rahimi BA, Thakkinstian A, White NJ, Sirivichayakul C, Dondorp AM, Chokejindachai W. Severe vivax malaria: a systematic review and meta-analysis of clinical studies since 1900. Malar J. 2014 Dec 8;13:481. doi: 10.1186/1475-2875-13-481. PMID 25486908
- [Background] Price RN, Tjitra E, Guerra CA, Yeung S, White NJ, Anstey NM. Vivax malaria: neglected and not benign. Am J Trop Med Hyg. 2007 Dec;77(6 Suppl):79-87. PMID 18165478
- [Background] Watson J, Taylor WRJ, Bancone G, Chu CS, Jittamala P, White NJ. Implications of current therapeutic restrictions for primaquine and tafenoquine in the radical cure of vivax malaria. PLoS Negl Trop Dis. 2018 Apr 20;12(4):e0006440. doi: 10.1371/journal.pntd.0006440. eCollection 2018 Apr. PMID 29677199
- [Background] Pybus BS, Marcsisin SR, Jin X, Deye G, Sousa JC, Li Q, Caridha D, Zeng Q, Reichard GA, Ockenhouse C, Bennett J, Walker LA, Ohrt C, Melendez V. The metabolism of primaquine to its active metabolite is dependent on CYP 2D6. Malar J. 2013 Jun 20;12:212. doi: 10.1186/1475-2875-12-212. PMID 23782898
- [Background] Bennett JW, Pybus BS, Yadava A, Tosh D, Sousa JC, McCarthy WF, Deye G, Melendez V, Ockenhouse CF. Primaquine failure and cytochrome P-450 2D6 in Plasmodium vivax malaria. N Engl J Med. 2013 Oct 3;369(14):1381-2. doi: 10.1056/NEJMc1301936. No abstract available. PMID 24088113
- [Background] Grabowsky M. The billion-dollar malaria moment. Nature. 2008 Feb 28;451(7182):1051-2. doi: 10.1038/4511051a. No abstract available. PMID 18305524
- [Background] Moorthy VS, Newman RD, Okwo-Bele JM. Malaria vaccine technology roadmap. Lancet. 2013 Nov 23;382(9906):1700-1. doi: 10.1016/S0140-6736(13)62238-2. Epub 2013 Nov 14. No abstract available. PMID 24239252
- [Background] Mueller I, Shakri AR, Chitnis CE. Development of vaccines for Plasmodium vivax malaria. Vaccine. 2015 Dec 22;33(52):7489-95. doi: 10.1016/j.vaccine.2015.09.060. Epub 2015 Oct 1. PMID 26428453
- [Background] Payne RO, Griffin PM, McCarthy JS, Draper SJ. Plasmodium vivax Controlled Human Malaria Infection - Progress and Prospects. Trends Parasitol. 2017 Feb;33(2):141-150. doi: 10.1016/j.pt.2016.11.001. Epub 2016 Dec 10. PMID 27956060
- [Background] Keith JA, Agostini Bigger L, Arthur PA, Maes E, Daems R. Delivering the promise of the Decade of Vaccines: opportunities and challenges in the development of high quality new vaccines. Vaccine. 2013 Apr 18;31 Suppl 2:B184-93. doi: 10.1016/j.vaccine.2012.12.032. PMID 23598480
- [Background] Pronker ES, Weenen TC, Commandeur H, Claassen EH, Osterhaus AD. Risk in vaccine research and development quantified. PLoS One. 2013;8(3):e57755. doi: 10.1371/journal.pone.0057755. Epub 2013 Mar 20. PMID 23526951
- [Background] Knezevic I, Moorthy V, Sheets R. WHO consultation on clinical evaluation of vaccines, 17-18 July 2014, WHO Headquarters, Geneva, Switzerland. Vaccine. 2015 Apr 21;33(17):1999-2003. doi: 10.1016/j.vaccine.2015.01.056. Epub 2015 Mar 4. PMID 25749249
- [Background] Stanisic DI, McCarthy JS, Good MF. Controlled Human Malaria Infection: Applications, Advances, and Challenges. Infect Immun. 2017 Dec 19;86(1):e00479-17. doi: 10.1128/IAI.00479-17. Print 2018 Jan. PMID 28923897
- [Background] Roestenberg M, Hoogerwerf MA, Ferreira DM, Mordmuller B, Yazdanbakhsh M. Experimental infection of human volunteers. Lancet Infect Dis. 2018 Oct;18(10):e312-e322. doi: 10.1016/S1473-3099(18)30177-4. Epub 2018 Jun 18. PMID 29891332
- [Background] Payne RO, Milne KH, Elias SC, Edwards NJ, Douglas AD, Brown RE, Silk SE, Biswas S, Miura K, Roberts R, Rampling TW, Venkatraman N, Hodgson SH, Labbe GM, Halstead FD, Poulton ID, Nugent FL, de Graaf H, Sukhtankar P, Williams NC, Ockenhouse CF, Kathcart AK, Qabar AN, Waters NC, Soisson LA, Birkett AJ, Cooke GS, Faust SN, Woods C, Ivinson K, McCarthy JS, Diggs CL, Vekemans J, Long CA, Hill AV, Lawrie AM, Dutta S, Draper SJ. Demonstration of the Blood-Stage Plasmodium falciparum Controlled Human Malaria Infection Model to Assess Efficacy of the P. falciparum Apical Membrane Antigen 1 Vaccine, FMP2.1/AS01. J Infect Dis. 2016 Jun 1;213(11):1743-51. doi: 10.1093/infdis/jiw039. Epub 2016 Feb 4. PMID 26908756
- [Background] McCarthy JS, Griffin PM, Sekuloski S, Bright AT, Rockett R, Looke D, Elliott S, Whiley D, Sloots T, Winzeler EA, Trenholme KR. Experimentally induced blood-stage Plasmodium vivax infection in healthy volunteers. J Infect Dis. 2013 Nov 15;208(10):1688-94. doi: 10.1093/infdis/jit394. Epub 2013 Aug 1. PMID 23908484
- [Background] Griffin P, Pasay C, Elliott S, Sekuloski S, Sikulu M, Hugo L, Khoury D, Cromer D, Davenport M, Sattabongkot J, Ivinson K, Ockenhouse C, McCarthy J. Safety and Reproducibility of a Clinical Trial System Using Induced Blood Stage Plasmodium vivax Infection and Its Potential as a Model to Evaluate Malaria Transmission. PLoS Negl Trop Dis. 2016 Dec 8;10(12):e0005139. doi: 10.1371/journal.pntd.0005139. eCollection 2016 Dec. PMID 27930652
- [Background] Collins KA, Wang CY, Adams M, Mitchell H, Robinson GJ, Rampton M, Elliott S, Odedra A, Khoury D, Ballard E, Shelper TB, Lucantoni L, Avery VM, Chalon S, Moehrle JJ, McCarthy JS. A Plasmodium vivax experimental human infection model for evaluating efficacy of interventions. J Clin Invest. 2020 Jun 1;130(6):2920-2927. doi: 10.1172/JCI134923. PMID 32045385
- [Background] Odedra A, Mudie K, Kennedy G, Watts RE, Rossignol E, Mitchell H, Gower J, Rebelo M, Pava Z, Pawliw R, Woolley S, Lalloo DG, Robinson G, Lynch S, Collins KA, Amante F, McCarthy J. Safety and feasibility of apheresis to harvest and concentrate parasites from subjects with induced blood stage Plasmodium vivax infection. Malar J. 2021 Jan 14;20(1):43. doi: 10.1186/s12936-021-03581-w. PMID 33446191
- [Background] Robinson S, Harris A, Atkinson S, Atterbury C, Bolton-Maggs P, Elliott C, Hawkins T, Hazra E, Howell C, New H, Shackleton T, Shreeve K, Taylor C. The administration of blood components: a British Society for Haematology Guideline. Transfus Med. 2018 Feb;28(1):3-21. doi: 10.1111/tme.12481. Epub 2017 Nov 6. No abstract available. PMID 29110357
- [Derived] Naemiratch B, Kulpijit N, Ruangkajorn S, Day NPJ, Prachumsri J, Cheah PY. Experiences, perceptions and ethical considerations of the malaria infection study in Thailand. BMC Med Ethics. 2025 Jan 28;26(1):14. doi: 10.1186/s12910-024-01160-7. PMID 39875955

DOCUMENTS (2):
  • Study Protocol (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05071079/Prot_002.pdf
  • Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT05071079/SAP_001.pdf